Trial Title: Cardiovascular Outcomes of an Adapted Evidence-Based Intervention for Rural

African Americans: Heart Matters Trial

**Internal Reference Number / Short title:** Heart Matters

ClinicalTrials.gov: NCT02707432

https://clinicaltrials.gov/ct2/show/NCT02707432?term=corbie&draw=2&rank=2

Other Study ID Number: UNC IRB - 13-2576

Chief Investigator: Giselle Corbie-Smith, MD, MSc

Department of Social Medicine

University of North Carolina at Chapel Hill

Investigators:

Leah Frerichs, PhD Tiffany L. Young, PhD Mysha Wynn, MA Shirley McFarlin, BA Crystal Cene, MD, MPH

Gaurav Dave, MD, DrPH, MPH

Funder: National Heart Lung and Blood Institute (Grant Number

1R01HL120690)

**Approval Date:** 2/25/20

No potential conflicts of interest.

# TABLE OF CONTENTS

| 1. | KEY | TRIAL CONTACTS | 4 |
|---|---|---|---|
| 2. | LAY | SUMMARY | 4 |
| 3. | SYN | NOPSIS | 5 |
| 4. | ABE | BREVIATIONS | 6 |
| 5. | BAC | CKGROUND AND RATIONALE | 6 |
| 6. | OB | JECTIVES AND OUTCOME MEASURES | 7 |
| 7. | TRI | AL DESIGN | 8 |
| 8. | PAF | RTICIPANT IDENTIFICATION | 8 |
| 8 | 3.1. | Trial Participants | 8 |
| 8 | 3.2. | Inclusion Criteria | 8 |
| 8 | 3.3. | Exclusion Criteria | 8 |
| 9. | TRI | AL PROCEDURES | 9 |
| Ś | 9.1. | Recruitment | |
| | 9.1 | 1.1 Organizational Recruitment | |
| c | 9.2. | Screening and Eligibility Assessment | |
| | 9.3. | Informed Consent | |
| | 9.4. | Randomization | |
| | 9.5. | Blinding and code-breaking | |
| | 9.6. | Baseline Assessments | |
| | 9.7. | Subsequent Visits | |
| | 9.7. | Sample Handling | |
| | 9.8.<br>9.9. | Early Discontinuation/Withdrawal of Participants | |
| | | Definition of End of Trial | |
| | | AFETY REPORTING | |
| 10. | | | |
| | | Adverse Event Definitions | |
| | | Adverse Events TATISTICS | |
| .11<br>ر | | | |
| | | Statistical Analysis Plan (SAP) | |
| | | Description of Statistical Methods | |
| | | Sample Size Determination | |
| | | Analysis Populations | |
| • | 115 | The Level of Statistical Significance | 13 |

| 11 | .6. Procedure for | Accounting for Missing, Unused, and Spurious Data | 13 |
|---|---|---|---|
| 11 | .7. Procedures fo | r Reporting any Deviation(s) from the Original Statistical P | lan 13 |
| 12. | DATA MANAGE | MENT | 13 |
| 12 | .1. Access to Data | a | 13 |
| 12 | 2. Data Recordin | g and Record Keeping | 13 |
| 13. | QUALITY ASSU | RANCE PROCEDURES | 13 |
| 13 | 3.1. Monitoring | | 14 |
| 13 | 3.2. Scientific Adviso | ory Board | 13 |
| 14. | PROTOCOL DE | VIATIONS | 14 |
| 15. | ETHICAL AND F | REGULATORY CONSIDERATIONS | 14 |
| 15 | i.1. Participant Co | nfidentiality | 14 |
| 15 | 5.2. Expenses and | Benefits | 14 |
| 16. | PUBLICATION F | POLICY | 14 |
| 17. | ARCHIVING | | 14 |
| 18. | REFERENCES. | | 15 |

#### 1 KEY TRIAL CONTACTS

| | RET TRIAL GORTAGIO |
|---|---|
| Chief Investigator | Giselle Corbie-Smith, MD, MSc<br>323 B MacNider<br>Dept Of Social Medicine<br>CB# 7240<br>Chapel Hill, NC 27599<br>(919) 966-7499<br>gcorbie@med.unc.edu |
| Funder(s) | National Heart, Lung, and Blood Institute (NHLBI) 5R01HL120690 |
| Clinical Trials Unit | Monica Coudurier Clinical Trials Project Manager UNC-CH Office of Clinical Trials 720 Martin Luther King, Jr. Blvd, CB 1651 Chapel Hill, NC 27599-1651 (919) 843-2333 Phone m_coudurier@unc.edu |
| Statistician | Feng-Chang Lin, PhD Associate Professor Department of Biostatistics 2nd floor, Brinkhous-Bullitt Building CB #7064 Chapel Hill, NC 27599 (919) 966-9431 flin@bios.unc.edu |
| Data Safety<br>Monitoring Board | |

#### 2 LAY SUMMARY

Cardiovascular disease (CVD) is the leading cause of death in the US, however African American residents of rural areas in the south and southeast regions have the highest prevalence of CVD of any group. African Americans carry a significant burden of CVD risk factors that often co-occur; this burden is amplified in rural communities. CVD disparities at the intersection of race and geography are driven by individual risk behaviors and complicated by factors such as limited access to quality healthcare, socio-economic inequities, limited healthcare infrastructure and environmental barriers to behavior change. Interventions to ameliorate CVD burden in rural African American communities will require placing the individual in the context of the larger community and taking advantage of new technologies to support behavior change. However, how best to integrate mobile technology into existing evidenced based interventions (EBIs) is still an emerging field and social and physical environmental factors important in rural communities are rarely considered in existing EBIs. The proposed study will address this gap in the literature by determining the feasibility and efficacy of adapting an EBI to consider the environment in important in rural African American communities and determining the acceptability of mobile technology in these communities to support behavior change. The proposed study is built on the

strong foundation of Project GRACE's 8-year history of designing and testing interventions using a community-based participatory research (CBPR) approach, and individual and collaborative expertise in community-based CVD outreach, service and research. We have developed a phased CBPR study with a long-term goal to reduce rates of CVD in Eastern NC. The overall objective of this proposal is to assess feasibility of implementing an EBI, adapted to the needs and interests of a rural community in order to plan a large scale study. To that end our specific aims are to 1) expand and sustain a Project GRACE CVD coalition of community and academic stakeholders to develop successful CVD risk prevention strategies in rural communities; 2) conduct a mixed-method community needs and assets assessment based on: a) assemble, review and assess existing sources of CVD data; b) identification of community strengths and resources using a web-based survey of community, faith based, social service and healthcare organizations; c) determine the acceptability of components of CVD risk reduction EBIs and community members' perceptions of possible targets for intervention using focus group interviews; d) determine specific family influences (barriers and facilitators) on acceptability of EBI acceptability: 3) adapt PREMIER, a multi-component EBI using intervention mapping; and 4) conduct a small-scale randomized control trial to assess a) efficacy; and, b) feasibility and adaption of implementing adapted PREMIER in rural settings.

#### 3 SYNOPSIS

| Trial Title | Cardiovascular Outcomes of an Adapted Evidence-Based Intervention for | | |
|---|---|---|---|
| | Rural African Americans: Heart Matters Trial | | |
| Internal ref. | Heart Matters | | |
| no. (or short | | | |
| title) | NOT2255422 | | |
| Trial | | NCT02707432 | |
| registration | Date of registration: March 14, 2016 https://clinicaltrials.gov/ct2/show/NCT02707432?term=corbie&draw=2&rank=2 | | |
| Funder | | | OIDIEQUIAW-ZQIAIIK-Z |
| | National Heart, Lung, and Blood Institute (NHLBI; 5R01HL120690) | | |
| Trial Design | Randomized, controlled trial | | |
| Trial<br>Participants | African American adults (21 years or older) with at least one risk factor for cardiovascular disease. | | |
| Sample Size | 140 | | |
| Planned Trial | Total length of the project is 1 | 8 months. Participant's in | volvement will be a |
| Period | 12-month intervention with a 6-month follow-up. | | |
| Planned<br>Recruitment<br>period | March 27, 2017 – February 28, 2019 | | |
| | Objectives | Outcome Measures | Timepoint(s) |
| Primary | To determine the effect of an adapted intervention, Heart Matters, on cardiovascular clinical outcomes. | Body weight | 6 months |
| Secondary | To determine the effect of Heart Matters on secondary cardiovascular clinical | Systolic and diastolic blood pressures | 6 months |

| | outcome | |
|---|---|---|
| Intervention(s) | rvention(s) Lifestyle modification consisting of interactive group and individual sessions targeting physical activity, weight loss, and nutrition. | |
| Comparator No comparator intervention due to delayed control des | | ue to delayed control design. |

#### 4 ABBREVIATIONS

| AE | Adverse event |
|-----|------------------------|
| PI | Principal Investigator |
| СТ | Clinical Trials |
| GCP | Good Clinical Practice |

#### 5 BACKGROUND AND RATIONALE

<u>Purpose:</u> To determine the effect of an adapted intervention, Heart Matters, on cardiovascular clinical outcomes.

Background: African Americans in the rural southeast are disproportionately affected by cardiovascular disease and associated risk factors. Despite evidence-based cardiovascular interventions targeting clinical or behavioral risk factors, geographic and racial disparities persist and continue to widen. Cardiovascular disease (CVD) is the leading cause of death in the United States (US) with an estimated 50% of individuals in the US expected to have CVD by 2030. African American residents in rural areas of the south and southeast (also called the "stroke belt") have the highest prevalence of CVD compared to other populations. Furthermore, CVD prevalence rates for residents of rural areas (13.1%) are higher compared to those in urban areas (11.2%) of the US. In the setting of geographic disparities, striking racial disparities in CVD risk factors, morbidity and mortality are exacerbated. African Americans are disproportionately affected by a higher burden of CVD risk factors: high blood pressure, diabetes, smoking, high cholesterol, and physical inactivity. This heightened risk is prevalent in both youth and older age groups and has increased over time. While CVD disparities at the intersection of race and geography are driven by a disproportionate burden of individual risk factors, racial disparities in rural settings are amplified by associated factors, such as limited access to quality healthcare services, socio-economic burden, dwindling resources, insufficient health infrastructure, and physical barriers to access to care. There are numerous evidence based interventions (EBIs) that have focused on reduction in CVD risk factors. These interventions have often focused on primary prevention of individual risk factors such as hypertension, diabetes, lipids, physical activity, and diet quality. Many of these have been developed in urban centers, and only a few have included participants that are reflective of geographic and racial disparities in CVD risk.

Given the burden of co-morbidities in rural African American populations, interventions targeting only one behavior or risk factor are likely to be less successful than those using intervention components and concepts impacting multiple behaviors. There is a need for culturally adapted interventions that address multiple behavioral risk factors for CVD. Using a Community-Based Participatory Research (CBPR) approach, our team adapted and will implement an EBI to improve cardiovascular risk in African Americans living in a rural underserved setting.

<u>Participants:</u> African Americans who reside in Edgecombe and Nash counties, aged 21 years or older, with at least one self-reported cardiovascular disease (CVD) risk factor.

Potential benefits for study participants include participation in long-term lifestyle modifications that may result in improved diet, nutrition, and physical activity patterns, which in turn should decrease blood pressure and lead to an overall reduction in cardiovascular and cancer morbidity.

Heart Matters Intervention: Heart Matters will use a lifestyle modification to reduce CVD risk factors and includes 26 interactive group sessions and 7 individual visit sessions over 12 months. Heart Matters lifestyle goals include: 1) reducing weight by 15 lbs. or another agreed upon goal, 2) limiting fat intake by consuming 20–50% or less of total calories from fat, 3) limiting daily sodium intake to 2300 mg or less, 4) accumulating 150 min of moderate-intensity exercise each week, 5) limiting alcohol intake; women are advised to consume no more than one alcoholic drink per day and men are advised to consume no more than two alcoholic drinks per day, and 6) diet and physical activity tracking.

Trained facilitators and co-facilitators will conduct 26 90-minute group sessions at each organizational site with 15–20 participants per group. Facilitators are members of the community who are teachers, coaches, or clergy members and have 30 min of group supervision of adherence to protocol for each session delivered. Co-facilitators are allied health professionals, such as nutritionists, nurses, and personal trainers who help deliver the educational content. All facilitators will participate in an extensive three-part training on intervention protocols and curriculum.

Participants will have seven 60-min individual sessions throughout the intervention. Individual sessions will be pre-scheduled and conducted via phone by the facilitator. Using motivational interviewing techniques, facilitators will discuss participant's progress and challenges to making behavior changes. Participants develop an individualized action plan at the first individual visit and this plan is revisited in subsequent individual visit sessions in an effort to track individual progress.

#### 6 OBJECTIVES AND OUTCOME MEASURES

| Objectives | Outcome Measures | Timepoint(s) of evaluation of this outcome measure (if applicable) |
|---|---|---|
| Primary Objective To determine the effect of an adapted intervention, Heart Matters, on body weight. | Body weight measured by Tanita WB-<br>800 Professional Digital Weight Scale | Body weight<br>measurement at<br>day 0 and 6<br>months after<br>baseline. |
| Secondary Objectives To determine the effect of an adapted intervention, Heart Matters, on cardiovascular clinical outcomes. | Systolic and diastolic blood pressures are measured by the Omron HEM907XL-Automatic Digital Blood Pressure Monitor. | All secondary outcomes are measured at day 0 and 6 months after baseline. |

#### 7 TRIAL DESIGN

Heart Matters is a community-based randomized trial comparing the effects of implementing the adapted lifestyle modification intervention on cardiovascular clinical outcomes among African American participants in rural eastern NC.

To implement Heart Matters, we will cluster individual participants within organizations that we recruit to participate in the study and be host sites for the intervention delivery. We will randomize organizations to 2 start times: Time 1 Heart Matters Intervention Group (immediately after baseline data collection) and Time 2 6 month-delay Heart Matters Intervention Group (6 months after baseline data collection). Randomization by organization will reduce the likelihood of data contamination given the fact that rural communities tend to be smaller and participants may be familiar with each other.

The flow of the participant is: 1. Screening at community organization and pre-intervention data collection. 2. Randomization of organizations to treatment group or 6 month delayed intervention control. 3. 6 month assessment data collection.

Data collection procedures: After the consent process, eligible individuals will complete the baseline data collection in a community setting. All data collection will be completed by trained research staff from the partner community organizations, James McFarlin Community Development, Inc and Project Momentum, Inc. Data collection will include biometric and biomarker data as well as self-report behavioral data. Trained research staff will collect biometrics such as weight, height, grip strength, and balance. Trained research staff who are registered nurses will collect blood pressure and hemoglobin A1c. Study staff will record the biometric data on paper forms which will be entered into REDCap, a secure web-based application for data management. For participants with life-threatening A1c levels, they will be immediately transported to emergency services, and adverse event data will be documented by research staff. The baseline questionnaire will include behavioral measures and structured questions on demographics (e.g. age, race, marital status, SES), health history, medications, CVD risk factors. Data collectors will enter data from the paper questionnaire forms into REDCap.

#### 8 PARTICIPANT IDENTIFICATION

### 8.1 Trial Participants

Participants with at least one risk factor for cardiovascular disease, living in one of two rural counties in eastern North Carolina, aged 21 years and older.

#### 8.2 Inclusion Criteria

- Participant is willing and able to give informed consent for participation in the trial.
- African American adults aged 21 years or above.
- Self-reported with at least one cardiovascular disease risk factor of pre-diabetes or diabetes, hypertension, obesity, family history of early CVD, or prior diagnosis of CVD

### 8.3 Exclusion Criteria

The participant may not enter the trial if ANY of the following apply:

Individuals who had significant cognitive impairment or unstable cardiovascular disease

Cognitive impairment that limits informed consent

### 9 TRIAL PROCEDURES

#### 9.1 Recruitment

## 9.1.1 Organizational Recruitment

We will recruit organizations to serve as recruitment and intervention sites from both counties (Edgecombe and Nash). We will invite potential organizations based on: (a) existing relationships through the Project GRACE consortium, (b) and a list of organizations beyond existing networks generated by our James McFarlin Community Development, Inc and Project Momentum, Inc collaborators. Knowing that CVD risk is high in older adult populations, the extended list will include senior health and civic organizations. Historically, faith based organizations reach a large segment of the minority community and are a trusted leader in the community. As a result, many organizations may be faith-based.

In addition to partnering for participant recruitment, organizations will be host sites for intervention delivery. We will use the following inclusion criteria to evaluate each organization: kitchen space with refrigerator, stove and/or microwave, contact person from each organization available to open and close the building, and layout of how the used space should look at the conclusion of use. We will base final inclusion criteria on if the site could host the intervention for all 12 months.Of the original list of criteria, we will identify sufficient sites to meet sample size needed.

# 9.1.2 Individual Participant Recruitment

Community-based recruiters at James McFarlin Community Development, Inc and Project Momentum, Inc will work with organizational leaders to hold recruitment events at each organization. Outreach to individuals will be based on recommendations from organizational leaders and will include direct outreach and information sessions at each organization, distributing written materials/flyers, recruiting at organizational events and exploring the social networks of initial recruits.

### 9.2 Screening and Eligibility Assessment

We will obtain verbal informed consent from potentially eligible participants for the initial screening during which individuals will provide identifiable information (e.g. contact information) and provide medical history to determine if eligible or excluded. No rescreening or protocol waivers will be permitted. Medical history interview will ask about cardiovascular disease risk factors (pre-diabetes or diabetes, hypertension, obesity, family history of early CVD, or prior diagnosis of CVD) and cognitive impairment.

### 9.3 Informed Consent

After the eligibility screening, we will obtain written informed consent for each eligible participant who decides to enroll in the study. Community partners at James McFarlin Community Development, Inc and Project Momentum, Inc will be responsible for enrolling participants into the study.

#### 9.4 Randomization

Participants in organizations will be randomized by a statistician into Time 1 (immediate intervention delivery after baseline data collection) and Time 2 (6 month delayed intervention delivery) under a matched pair in order to balance the sample size between Arm 1 and 2. Organizations will be paired based on the number of participants, and then randomly assigned one organization from each pair to each arm.

# 9.5 Blinding and code-breaking

There is no blinding or code-breaking in this trial.

#### 9.6 Baseline Assessments

Immediately following the consent process, eligible individuals will complete the baseline data collection in a community setting. All data collection is completed by trained research staff from the partner community organizations, James McFarlin Community Development, Inc and Project Momentum, Inc. Data collection will include biometric and biomarker data as well as self-report behavioral data. Trained research staff will collect weight. Trained research staff who are registered nurses will collect blood pressure and hemoglobin A1c. Study staff will record the biometric data on paper forms which will be entered into REDCap, a secure web-based application for data management. For participants with life-threatening A1c levels, they will be immediately transported to emergency services, and adverse event data will be documented by James McFarlin Community Development, Inc and Project Momentum, Inc research staff.

Trained data collectors will conduct the structured survey. The baseline questionnaire will include behavioral measures and structured questions on demographics (e.g. age, race, marital status, SES), health history, medications, CVD risk factors. Data collectors will enter data from the paper questionnaire forms into REDCap.

### 9.7 Subsequent Visits

Data collection occurs at baseline and at each 6 month interval for 18 months.

# 9.8 Sample Handling

All samples for A1C will be disposed as biohazard material immediately after collection, reading, and recording is complete.

### 9.9 Early Discontinuation/Withdrawal of Participants

During the course of the trial a participant may choose to withdraw early from the trial at any time. This may happen for a number of reasons, including but not limited to:

- The occurrence of what the participant perceives as an intolerable adverse event.
- Inability to comply with trial procedures
- Participant decision due to circumstances outside of trial.

Participants may have the following two options for withdrawal;

- Participants can withdraw from the study but permit data and samples obtained up until
  the point of withdrawal to be retained for use in the study analysis. No further data or
  samples would be collected after withdrawal.
- 2) Participants can withdraw completely from the study and withdraw the data and samples collected up until the point of withdrawal. The data and samples already collected would not be used in the final study analysis. (Any limits to this type of withdrawal where, for example analysis of their data or samples has already been integrated into interim results or dose escalation decisions etc. should be explained in the participant information sheet).

In addition, the Investigator may discontinue a participant from the trial treatment at any time if the Investigator considers it necessary for any reason including, but not limited to:

- Ineligibility (either arising during the trial or retrospectively having been overlooked at screening)
- An adverse event which requires discontinuation of the trial or results in inability to continue to comply with trial procedures

#### 9.10 Definition of End of Trial

The end of trial is the point at which all the data has been collected and entered and no participant contact is needed.

#### 10 SAFETY REPORTING

Safety reporting will be addressed during routing study team meetings and additional as needed meetings or communication. The PI and study coordinator will report any safety issues to the IRB. The IRB will be notified of any safety issues that necessitate reporting and possible protocol changes. Progress reports will be provided to the IRB at least annually, or as requested. All unanticipated problems or serious adverse events involving risk to human subjects will be reported. All collaborators, students, and employees assisting in this research study will be informed about these obligations.

### **10.1 Adverse Event Definitions**

| Adverse Event (AE) | Any untoward medical occurrence in a participant to whom a medicinal product has been administered, including occurrences which are not necessarily caused by or related to that product. |
|---|---|
| Serious Adverse Event (SAE) | A serious adverse event is any untoward medical occurrence that: • results in death • is life-threatening • requires inpatient hospitalisation or prolongation of existing hospitalisation • results in persistent or significant disability/incapacity • consists of a congenital anomaly or birth defect*. |

Other 'important medical events' may also be considered a serious adverse event when, based upon appropriate medical judgement, the event may jeopardise the participant and may require medical or surgical intervention to prevent one of the outcomes listed above.

#### 10.2 Adverse Events

In the event of an adverse event, the PI and study team will work with the IRB to determine a protocol for handling AE that may occur during the course of data collection and the intervention. Facilitators and data collectors will be trained to follow protocol procedures and report any AE to the primary investigator immediately.

### 11 STATISTICS

## 11.1 Statistical Analysis Plan (SAP)

The plan for the statistical analysis of the trial are outlined below. There is not a separate SAP document in use for the trial.

# 11.2 Description of Statistical Methods

Demographics and clinical measures will be described using means, standard deviations, frequencies, and percentages. T-tests will be used to compare group level characteristics of continuous variables. Pearson Chi-square tests will be used to compare categorical group comparisons. Treatment effects from baseline to 6 months post intervention will be analyzed using linear mixed effects models. Least square means differences will be used by finding the differences between baseline and 6-month outcomes, as well as differences in groups with corresponding 95% confidence intervals. Models will be adjusted for age, blood pressure medications, and cluster. All of the analysis will be implemented using SAS 9.4 (Cary, NC).

### 11.3 Sample Size Determination

Sample size for Heart Matters was calculated on the basis of observing a 1.8 kg difference (SD = 3.2) in the primary outcome – weight change – between two intervention groups from baseline to 6 months. We determined a sample of 102 would allow us to detect a 1.8 kg difference (SD = 3.2) in weight change between intervention and control groups, with 80% power and an  $\alpha$  of 0.05. Accounting for attrition and intra-class correlation, due to a clustered randomized delayed intervention design, we plan to enroll 120 participants.

### 11.4 Analysis Populations

We will implement Heart Matters in Edgecombe and Nash counties; two counties in eastern North Carolina that are considered rural by urbanized area definitions with respective populations of 54,150 and 93,919. The two counties share one urbanized area, the city of Rocky Mount. Both have had a large prevalence of African Americans (56.7 and 40% of population, respectively) that experience significant health disparities with respect to cardiovascular disease. The sample is recruited through community organizations and

thus not considered a randomly selected sample representative of populations.

# 11.5 The Level of Statistical Significance

A p-value smaller than 0.05 will be considered statistically significant.

### 11.6 Procedure for Accounting for Missing, Unused, and Spurious Data

For all measures, scores will be calculated if an individual answered at least 60% of the items of a given measure. If an individual answered less than 60% of items, the data will be treated as missing for that measure only.

**11.7 Procedures for Reporting any Deviation(s) from the Original Statistical Plan** Any deviations from the original statistical analysis plan will be reported in publications.

# 12 DATA MANAGEMENT

Data collection will include biometric and biomarker data as well as self-report behavioral data. Hard copy files of data will be retained in locked containers in locked rooms where approved study staff will have access. Data will be entered in REDCap, a secure web-based application for data management. All export of data from REDCap will adhere to university protocols to ensure data is safely stored on university approved servers.

#### 12.1 Access to Data

Direct access will be granted to authorized representatives from the Sponsor, host institution and the regulatory authorities to permit trial-related monitoring, audits and inspections.

### 12.2 Data Recording and Record Keeping

Trained research staff will collect weight and other data collection except trained research staff who are registered nurses will collect blood pressure and hemoglobin A1c. Study staff will record the biometric data on paper forms, which will be entered into REDCap, a secure web-based application for data management. REDCap provides timestamped tracking to allow for an audit trail of all revisions to database codebook and data itself. Any quality assurance reviews and corrections to data entry will be tracked through REDCap.

Hard copy files will be stored at UNC. The participants will be identified by a unique trial specific number and/or code in any database. The name and any other identifying detail will NOT be included in any trial data electronic file. Informed consent documents and a document linking file that links participant ID to their name will be stored separately from all data.

### 13 QUALITY ASSURANCE PROCEDURES

### 13.1 Monitoring

Weekly meetings will be conducted with the team members during all stages of the study to review progress to date, any protocol deviations, data management, safety monitoring, and compliance.

### 13.2 Scientific Advisory Board

The Scientific Advisory Board will be comprised of PI, Co-Investigator, Project Manager, Biostatistician from the study two and 2 outside experts. The study team will provide a report to the scientific advisory board annually, and the board will discuss and make recommendations to support completion of scientific aims. As this will be a minimal risk study, this oversight is sufficient.

#### 14 PROTOCOL DEVIATIONS

A trial related deviation is a departure from the ethically approved trial protocol or other trial document or process (e.g. consent process) or any applicable regulatory requirements. Any deviations from the protocol will be documented in a protocol deviation form and filed in the trial master file. The protocol deviations and completed forms will be presented to the PI and study team by the project coordinator during weekly meetings. The review will ensure any repetitive or single, but significant deviations be escalated to the IRB for assessment of whether a non-compliance /deviation may be a potential Serious Breach and determine any necessary response.

#### 15 ETHICAL AND REGULATORY CONSIDERATIONS

### 15.1 Participant Confidentiality

To track participant outcomes across time while maintaining confidentiality, ID numbers will be used. A separate linking file will be maintained linking the IDs to the respondents' names. The surveys will be conducted using the mobile REDCap database, a password protected, firewalled database only accessible to the research team. Data will be collected using RedCap app. In case of computer problems, we will have paper copies of surveys available. All paper documentation will be maintained in locked files at UNC.

## 15.2 Expenses and Benefits

Participants will receive \$195 in compensation for participation in data collection and intervention session attendance: \$5 eligibility screening, \$25 for baseline data collection, \$15 for 6 month data collection, \$20 for 12 month data collection, and \$20 for 18 month data collection. Throughout the intervention, participants will receive a \$15 cash incentive for attendance at Group Sessions 4, 8, 12, 16, 20, 24, and \$20 at session 26.

#### 16 PUBLICATION POLICY

The study PI is responsible for intellectual content on publications from the dataset collected for this study. Study PI should determine appropriate authorship and acknowledgements for all scientific publications. Institutional and funder policies should be adhered to. NHLBI should be acknowledged in all publications.

## 17 ARCHIVING

6 months after the main study outcomes paper is published, de-identified dataset will be available per institutional and federal guidelines. Data will be destroyed five years after the study

publications are complete. For electronic data, we will follow accepted techniques to permanently delete files. This will include destruction of linkage files, transcriptions, data files, web-based database files, digital interviews and all other electronic files. All paper files will be shredded at that time.

#### 18 REFERENCES

ACSM-American College of Sports Medicine. *ACSM's Guidelines for Exercise Testing and Prescription*. Fifth Edition. Media, PA: Williams and Wilkins, 1995.

Aickin M, Ritenbaugh C. A criterion for the adequacy of sample size calculations based on a simple model when a complex model will be used for the analysis. *Control Clin Trials* 1991; 12:560-565.

Ainsworth BE, Keenan NL, Strogatz DS, Garrett JM, James SA: Physical activity and hypertension in black adults: The Pitt County Study. *Am J Public Health* 1991; 81:1477-1479.

Alderman MH, Cohen H, Madhaven S. Dietary sodium intake and mortality: the National Health and Nutrition Examination Survey. *Lancet* 1998; 351:781-5.

Alderman MH, Madvan S, Cohen H, Sealey JE, Laragh JH. Low urinary sodium is associated with greater risk of myocardial infarction among treated hypertensive men. *Hypertension* 1995; 25:1144-1152.

Ammerman A, Caggiula A, Elmer PJ, Kris-Etherton P, Keyserling T, Keyserling T, Lewis C, Luepker R, Pearson T, Schucker B Shannon B, Simpson Jr RJ, Watson J. Putting medical practice guidelines into practice: The cholesterol model. *Am J Prev Med* 1994; 10:209-216.

Appel LJ, Espeland MA, Dorshenko, Bottom J, Lacy CR, Wilson AC, *et al.* Reduced sodium intake as a means to control high blood pressure in older-aged adults: Results from the Trial of Nonpharmacologic Interventions in the Elderly (TONE). *Can J Cardiol* 1997a; 13:206B.

Appel LJ, Espeland M, Whelton PK, Dolecek T, Kumanyika S, Applegate WB, *et al.* Trial of Nonpharmacologic Intervention in the Elderly (TONE): Design and rationale of a blood pressure control trial. *Ann Epidemiol* 1995; 5:119-129.

Appel LJ, Moore TJ, Obarzanek E, Vollmer WM, Svetkey LP, Sacks FM, et al. A clinical trial of the effects of dietary patterns on blood pressure. *N Engl J Med* 1997b; 336:1117-1124.

Arroll B, Beaglehole R. Does physical activity lower blood pressure: A critical review of the clinical trials. *J Clin Epidemiol* 1992; 45:439-447.

Ascherio A, Rimm EB, Hernan MA, Giovannucci EL, Kawachi I, Stampfer MJ, Willett WC. Intake of potassium, magnesium, calcium, and fiber and risk of stroke among US men. *Circulation* 1998; 98:1198- 204.

Bandura A. Social Foundations of Thought and Action. A Social Cognitive Theory. Englewood Cliffs: Prentice Hall, 1986.

Blair SN, Applegate WB, Dunn AL, Ettinger WH, Haskell WL, King AC, Morgan TM, Shih JH, Simons- Morton DG. Activity Counseling Trial (ACT): Rationale, design, and methods. *Med Sci Sports Exerc* 1998; 30:1097-1106.

Blair SN, Haskell WL, Po H, Paffenbarger Jr RS, Vranizan KM, Farquhar JW, Wood PD. Assessment of habitual physical activity methodology by a seven-day recall in a community survey and controlled experiments. *Am J Epidemiol* 1986; 122:794-804.

Bohn MJ, Babor TF, Kranzler HR. The Alcohol Use Disorders Identification Test (AUDIT): Validation of a screening instrument for use in medical settings. *J Stud Alcohol* 1995; 56:423-432.

Borg GAV. Psychological bases of perceived exertion. *Med Sci Sports Exerc*; 1982; 14:377-381.

Braith RW, Pollock ML, Lownthal DT, Graves JE, Limacher MC. Moderate and high-intensity exercise lowers blood pressure in normotensive subjects 60 to 79 years of age. *Am J Cardiol* 1994;73:1124-1128.

Budd MA, Gruman JC. Behavioral medicine: Taking its place in the mainstream of primary care. *HMO Pract* 1995; 9(2):51-52.

Burnes H. Personal health improvement program. HMO Pract 1995; 9:59-60.

Burt VL, Whelton P, Roccella EJ, Brown C, Cutler JA, Higgins M, *et al.* Prevalence of hypertension in the U.S. adult population: Results from the Third National Health and Nutrition Examination Survey, 1988-1991. *Hypertension* 1995; 25:305-313.

Cohen S, Kamarck R, Mermelstein R. A global measure of perceived stress. *J Health Soc Behav*, 1983;24:385-396

Cohen, S, Williamson, GM Perceived stress in a probability sample of the United States. In S. Spacapan & S. Oskamp (eds.), The Social Psychology of Health. Newbury Park, CA: Sage, 1988.

Collins R, Peto R, MacMahon S, Hebert P, Fiebach NH, Eberlein KA, Godwin J, Qizilbash N, Taylor JO, Hennekens C: Blood pressure, stroke, and coronary heart disease. Part 2, short-term reductions in blood pressure: overview of randomised drug trials in their epidemiological context. *Lancet* 1990; 335:827-838.

Coresh J, Mead L, Levine DM, Klag MJ. Increased cardiovascular disease risk in treated hypertensive men. AHA 66th Scientific Sessions. *Circulation* 1993; 88:I-124 [abstract].

Cushman WC, Cutler JA, Hanna E, Bingham SF, Follmann D, Harford T, Dubbert P, Allender S, *et al.* The Prevention and Treatment of Hypertension Study (PATHS) Effects of an Alcohol Treatment Program on Blood Pressure. *Arch Intern Med* 1998; 158:1197-1207

Cutler JA, Follmann, Allender PS. Randomized trials of sodium reduction: an overview. *Am J Clin Nutr.* 1997; 65:643S-651S.

Dunn AL, Marcus BH, Kampert JB, Garcia ME, Kohl HW, Blair SN. Reduction in cardiovascular disease risk factors: 6-month results from Project Active. *Prev Med* 1997; 26:883-892.

Elliott P, Stamler J, Nichols R, Dyer A, Stamler R, Kesteloot H, *et al.* Intersalt revisited: further analyses of 24 hour sodium excretion and blood pressure variation within and across populations. *BMJ* 1996; 312:1249-53.

Elmer PJ, for the DELTA Investigators. Effects of a step1 diet and a high monounsaturated (MUFA) fat diet on hemostatic factors in individuals with markers for insulin resistance. *FASEB J* 1996a; 10:2667.

Elmer PJ, for the DELTA Investigators. Effects of altering dietary fat-total & fatty acids on hemostatic factors. *Circulation* 1996b; 94:SI690.

Elmer PJ, Fosdick L, Tharp TM, Smith SA, Laing B, Potter J. Feasibility of increasing vegetable & fruit intake for colon cancer prevention. *Cancer Epidemiol Biomarkers Prev* 1995b; 4:183.

Elmer PJ, Fosdick L, Tharp T, Smith S, Laing B, Potter J. Increased vegetable & fruit intake for cardiovascular disease prevention. *Circulation* 1994; 90:2:I-74.

Elmer PJ, Grimm RH, Flack J, Laing B. Dietary sodium reduction for hypertension prevention and treatment in clinical and community settings. *Hypertension* 1991; 14:98-108.

Elmer PJ, Grimm R, Laing B, Grandits G, Svendsen K, Van Heel N, *et al.* Lifestyle intervention of the Treatment of Mild Hypertension study (TOMHS). *Prev Med* 1995a; 24:378-388.

Fagard RH. Physical fitness and blood pressure. J Hypertens 1993; 11:S47-S52.

Fagard RH. Prescription and results of physical activity. *J Cardiovasc Pharmacol* 1995; 25:S20-S27.

Frost CD, Law MR, Wald NJ. By how much does dietary salt reduction lower blood pressure? II. Analysis of observational data within populations. *BMJ* 1991; 302:815-818.

Gill TM, Feinstein AR. A critical appraisal of the quality of quality-of-life measurements. *JAMA* 1994; 272(8):619-626

Gillman MW, Cupples LA, Gagnon D, Posner BM, Ellison RC, Castelli WP, Wolf PA. Protective effect of fruits and vegetables on development of stroke in men. *JAMA* 1995; 273(14):1113-1117.

Grimm RH, Grandits GA, Elmer PJ. The Treatment of Mild Hypertension Study: final results of quality of life measures with diet and drug treatment of mild hypertension. *Arch Intern Med* 1997:157:638-648

Grimm RH, Neaton JD, Elmer PJ, Svendsen KH, Levin J, Segal M, Holland L, Witte LJ, Clearman DR, Kofron P, LaBounty RK, Crow R, Prineas RJ. The influence of oral potassium chloride on blood pressure in hypertensive men on a low-sodium diet. *N Engl J Med* 1990; 322:569-574.

Hagberg JM, Montain SJ, Martin WH, Ehsani AA. Effect of exercise training in 60- to 69-year-old persons with essential hypertension. *Am J Cardiol* 1989; 64:348-353.

Harris JR, Gordon RL, White KE, Strange PV, Harper SM. Prevention and managed care: Opportunities for managed care organizations, purchasers of health care, and public health agencies. *HMO Pract* 1996; 10:24-29.

Holm, S. A simple sequentially rejective multiple test procedure. *Scand. J. Statistics* 1979; 6:65-70.

INTERSALT Cooperative Research Group. INTERSALT: an international study of electrolyte excretion and blood pressure. Results for 24 hour urinary sodium and potassium excretion. *BMJ* 1988; 297:319- 328.

Jeffery RW. Weight management and hypertension. Ann Behav Med 1991; 13:18-22.

JNC V-Joint National Committee on Detection, Evaluation, and Treatment of High Blood Pressure: The Fifth report of the Joint National Committee on Detection, Evaluation, and Treatment of High Blood Pressure. Arch Intern Med 1993; 153:154-183.

JNC VI-Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. The Sixth Report of the Joint National Committee on the Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Arch Intern Med 1997; 157:2413-2446.

Kelley G, McClellan P. Antihypertensive effects of aerobic exercise. A brief meta-analytic review of randomized controlled trials. *Am J Hypertens* 1994; 7:115-119.

Kelley G, Tran ZV. Aerobic exercise and normotensive adults: a meta-analysis. . *Med Sci Sports Exerc.* 1995; 27:1371-1377.

Khaw KT, Barrett-Connor E. Dietary potassium and stroke-associated mortality. *N Engl J Med* 1987; 316:235-240.

King AC, Haskell WL, Taylor CB, Kraemer HC, DeBusk RF. Group vs home-based exercise training in healthy older men and women. *JAMA* 1991; 266:1535-1542.

King AC, Taylor CB, Haskell WL, DeBusk RF. Identifying strategies for increasing employee physical activity levels: Findings from the Stanford/Lockheed exercise survey. *Health Educ Q* 1990; 17:269-285.

Klatsky AL, Friedman GD, Siegelaub AB, Gerard MJ. Alcohol consumption and blood pressure. *N Engl J Med* 1977; 296:1194-1200.

Kuczmarski RJ, Flegal KM, Campbell SM, Johnson CL. Increasing prevalence of overweight among U.S. adults: The National Health and Nutrition Examination Surveys, 1960 to 1991. *JAMA* 1994; 272:206-211.

Kumanyika S, Herbert PR, Cutler JA, Lasser VI, Sugars CP, Steffen-Batey L, *et al.* Feasibility and efficacy of sodium reduction in the Trials of Hypertension Prevention, Phase I. *Hypertension* 1993; 22:502-512.

Lan, K.K.G. and DeMets, D.L. (1983). Discrete sequential boundaries for clinical trials. *Biometrika* 70, 659-663.

Lan, K.K.G., Simon, R., and Halperin, M. (1982). Stochastically curtailed tests in long term clinical trials. *Communications in Statistics-Sequential Analysis* 1(3), 207-219.

Lan, K.K.G. and Wittes, J. (1988). The B-value; a tool for monitoring data. *Biometrics* 44, 579-585.

Lasser VI, Raczynski JM, Stevens VJ, Mattfeldt-Beman MK, Kumanyika S, Evans M, Danielson E, Dalcin A, Batey DM, Belden LK, Brewer AA. Trials of Hypertension Prevention, Phase II: Structure and content of the weight loss and dietary sodium reduction interventions. *Ann Epidemiol* 1995; 5: 156- 164.

Law MR, Frost CD, Wald NJ. By how much does dietary salt reduction lower blood pressure? I. Analysis of observational data among populations. *BMJ* 1991; 302:811-815.

Lorig K. Arthritis self-help course. HMO Pract 1995; 9:60-61.

Lorig KR, Mazonson PD, Holman HR. Evidence suggesting that health education for self-management in patients with chronic arthritis has sustained benefits while reducing health care costs. *Arthritis Rheum* 1993; 36:439-446.

MacMahon S. Alcohol consumption and hypertension. *Hypertension* 1987; 9:111-121.

MacMahon S, Peto R, Cutler J, Collins R, Sorlie P, Neaton J, Abbott R, Goodwin J, Dyer A, Stamler J. Blood pressure, stroke, and coronary heart disease. Part 1, prolonged differences in blood pressure: prospective observational studies corrected for the regression dilution bias. *Lancet* 1990; 335:765-774.

Mant D. Effectiveness of dietary intervention in general practice. *Am J Clin Nutr* 1997; 65(suppl):1933S-1938S.

Marcus BH, Banspach SW, Lefebvre RC, Rossi JS, Carleton RA, Abrams DB. Using the stages of change model to increase the adoption of physical activity among community participants. *Am J Health Promot* 1992; 6:424-429.

Marlatt GA, Gordon JR (Eds.). *Relapse Prevention: Maintenance Strategies in the Treatment of Addictive Behaviors.* New York: Guilford Press, 1985.

McAfee T, Wilson J, Dacey S, Sofian N, Curry S, Wagener B. Awaking the sleeping giant: Mainstreaming efforts to decrease tobacco use in an HMO. *HMO Pract* 1995; 9:138-143.

Miller NH, Warren D, Myers D. Home-based cardiac rehabilitation and lifestyle modification: The MULTIFIT model. *Journal Cardiovasc Nurs* 1996; 11:76-87.

Miller WR, Rollnick S. *Motivational Interviewing: Preparing People to Change Addictive Behavior*. New York: The Guilford Press, 1991.

Neaton J, Grimm R, Prineas R, Stamler J, Grandits G, Elmer PJ, Cutler J, Flack J, Schoenberger, J, McDonald R, Lewis C, Liebson P, for the Treatment of Mild Hypertension

Research Group. Treatment of Mild Hypertension Study (TOMHS): Final results. *JAMA* 1993; 270(6):713-724.

NHLBI (National Heart, Lung, and Blood Institute). Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults - The Evidence Report. *Obesity Research* 1998 Sep; 6 Suppl:51S-209S

NIH Consensus Conference. Physical activity and cardiovascular health. *JAMA* 1996; 276:241-246.

O'Brien, P.C. and Fleming, T.R. (1979). A multiple testing procedure for clinical trials. *Biometrics* 33, 549-556.

Pate RR, Pratt M, Blair SN, Haskell WL, Macera CA, Bouchard C, Buchner D, *et al.* Physical activity and public health. A recommendation from the Centers for Disease Control and the American College of Sports Medicine. *JAMA* 1995; 273:402-407.

Plewis I. Analysing Change Chichester UK: John Wiley & Sons, 1985.

Pollock ML, Carroll JF, Graves JE, Leggett SH, Braith RW, Limacher M, Hagberg JM. Injuries and adherence to walk/jog and resistance training programs in the elderly. *Med Sci Sports Exerc* 1991; 23:1194-1200.

Proschan MA. A multiple comparison procedure for three- and four-armed controlled clinical trials. *Stat Med* 1999; 18:787-798.

Prochaska JO, DiClemente CC. Stages and process of self-change in smoking: Towards an integrative model of change. *J Consult Clin Psychol* 1983; 51:390-395.

Psaty BM, Heckbert SR, Koepsell TD, Siscovick DS, Raghunathan TE, Weiss NS, *et al.* The risk of myocardial infarction associated with antihypertensive drug therapies. *JAMA* 1995; 274:620-655.

Puddey IB, Beilin LJ, Vandongen R. Regular alcohol use raises blood pressure in treated hypertensive subjects. *Lancet* 1987; 1:647-651.

Puddey IB, Beilin LJ, Vandongen R, Rouse IL, Rogers P. Evidence for a direct effect of alcohol consumption on blood pressure in normotensive men: A randomized controlled trial. *Hypertension* 1985; 7:707-713.

Reaven PD, Barrett-Connor E, Edelstein S. Relation between leisure time physical activity and blood pressure in older women. *Circulation* 1991; 83:559-565.

Roman O, Camuzzi AL, Villalon E, Klenner C. Physical training program in arterial hypertension. A long-term prospective follow-up. *Cardiology* 1981; 67:230-243.

Rose G, McCartney P, and Reid DD. Self-administration of a questionnaire on chest pain and intermittent claudication. *Br J Prev Soc Med* 1977; 31:42-48.

Sacks FM, Obarzanek E, Windhauser MM, Svetkey LP, Vollmer WM, *et al.* Rationale and design of the Dietary Approaches to Stop Hypertension trial (DASH). *Ann Epidemiol* 1995; 5:108-118.

Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader. The development of scales to measure social support for diet and exercise behaviors. *Prev Med* 1987;16:825-836.

Sallis JF, Haskell WL, Wood PD, Fortmann SP, Rogers T, Blair SN, Paffenbarger Jr RS. Physical activity assessment methodology in the Five-City Project. *Am J Epidemiol* 1985; 121:91-106.

Sallis JF, Hovell MF, Hofstetter CR, Barrington E. Explanation of vigorous physical activity during two years using social learning variables. *Soc Sci Med* 1992;34:25-32.

Sallis JF, Pinski RB, Grossman RM, Patterson TL, Nader PR. The development of self-efficacy scales for health-related diet and exercise behaviors. *Health Education Research*, 1988;3:283-292.

Satterfield S, Cutler JA, Langford HG, Applegate WB, Borhani NO, Brittain E, Cohen JD, Kuller LH, Lasser NL, Oberman A, Rosner B, Taylor JO, Vogt TM, Walker G, Whelton PK. Trials of Hypertension Prevention: Phase I design. *Ann Epidemiol* 1991; 1:455-471.

SHEP Cooperative Research Group. Prevention of stroke by antihypertensive drug treatment of older persons with isolated systolic hypertension: Final results of the Systolic Hypertension in the Elderly Program (SHEP). *JAMA* 1991; 265:3255-3264.

Sidney S, Jacobs DR Jr, Haskell WL, Armstrong MA, Dimicco A, Oberman A, Savage PJ, Slattery ML, Sternfeld B, VanHorn L. Comparisons of two methods of assessing physical activity in the Coronary Artery Risk Development in Young Adults (CARDIA) Study. *Am J Epidemiol* 1991; 133:1231-1245.

Smiciklas-Wright HA, Mitchell MS, Norton LD, Derr JA. Interviewer reliability of nutrient intake data from 24-hour recalls collected using the Minnesota Nutrition Data System (NDS). *J Am Diet Assoc* 1991; 91:A28.

Solberg LI, Kottke TE, Brekke ML, Calomeni CA, Conn SA, Davidson G. Using continuous quality improvement to increase preventive services in clinical practice-going beyond guidelines. *Prev Med* 1996; 25:259-267.

Staessen J, Fagard R, Lijnen P, Amery A. Body weight, sodium intake, and blood pressure. *J Hypertens.* 1989; 7:S19-S23.

Stamler J. Epidemiologic findings on body mass and blood pressure in adults. *Ann Epidemiol* 1991; 1:347-362

Stamler J, Stamler R, Neaton JD. Blood pressure, systolic and diastolic, and cardiovascular risks: U.S. population data. *Arch Intern Med* 1993;153:598-615

Stamler R, Stamler J, Gosch FC, Civinelli J, Fishman J, McKeever P, McDonald A, Dyer AR. Primary prevention of hypertension by nutritional-hygienic means. *JAMA* 1989; 262:1801-1807.

Stamler R, Stamler J, Grimm R, Gosch FC, Elmer P, Dyer A, Berman R, Fishman J, Van Heel N, Civinelli J, McDonald A. Nutritional therapy for high blood pressure. Final report of a four-year randomized control trial--The Hypertension Control Program. *JAMA* 1987; 257:1484-1491.

Steinmetz KA, Potter JD. Vegetables and fruit and cancer prevention: A review. *J Am Diet Assoc* 1996; 96:1027-1039.

Stevens VJ, Corrigan SA, Obarzanek E, Bernauer E, Cook NR, Hebert P, Mattfeldt-Beman M, Oberman A, Sugars C, Dalcin AT, Whelton PK, for the TOHP Collaborative Research Group. Weight loss intervention in Phase I of the Trials of Hypertension Prevention. *Arch Intern Med* 1993; 153:849-858.

Stevens VJ, Rossner J, Greenlick MR, Stevens N, Frankel HM, Craddick S. Freedom from Fat: A contemporary multicomponent weight loss program for the general population of obese adults. *J Am Diet Assoc* 1989; 89:1254-8.

Stunkard AJ, Sorensen R, Schulsinger F. Use of the Danish Adoption Register for the study of obesity and thinness. Genetics of Neurological and Psychiatric Disorders, 1983;115-120.

Svetkey LP, Simons-Morton D, Vollmer WM, Appel LJ, Conlin PR, Ryan DH, Ard J, Kennedy BM; for the DASH Research Group. Effects of Dietary Patterns on Blood Pressure: Subgroup Analysis of the Dietary Approaches to Stop Hypertension (DASH) Randomized Clinical Trial. *Arch Intern Med* 1999; 159:285-293

TACP-Technology Assessment Conference Panel. Methods for voluntary weight loss and control: Technology Assessment Conference statement. *Ann Intern Med* 1992; 116:942-949.

TOHP1-The Trials of Hypertension Prevention Collaborative Research Group. The effects of nonpharmacologic interventions on blood pressure of persons with high-normal levels: Results of the Trials of Hypertension Prevention, Phase I. *JAMA* 1992; 267:1213-1220.

TOHP2-The Trials of Hypertension Prevention Collaborative Research Group. Effects of weight loss and sodium reduction intervention on blood pressure and hypertension incidence in overweight people with high-normal blood pressure: The Trials of Hypertension Prevention, Phase II. *Arch Intern Med* 1997; 157:657-667.

TOMHS-The Treatment of Mild Hypertension Research Group. The Treatment of Mild Hypertension Study: A randomized, placebo-controlled trial of nutritional-hygienic regimen along with various drug monotherapies. *Arch Intern Med* 1991; 151:1413-1423.

Tulkin SR. Pain management program. HMO Pract 1995; 9:57-58.

Tuomilehto J, Marti B, Salonen JT, Virtala E, Lahti T, Puska P. Leisure-time physical activity is inversely related to risk factors for coronary heart disease in middle-aged Finnish men. *Eur Heart J* 1987; 8:1047-1055.

USDHHS-U.S. US Department of Health and Human Services. *Physical Activity and Health: A Report of the Surgeon General.* Atlanta, GA: US Department of Health and Human Services, Centers for Disease Control and Prevention, National Center for Chronic Disease Prevention and Health Promotion, 1996.

Van Horn LV, Dolecek TA, Grandits GA, Skweres L. Adherence to dietary recommendations in the special intervention group in the Multiple Risk Factor Intervention

Trial. Am J Clin Nutr 1997; 65(suppl):289S-304S.

Ware JE. *SF-36 Health Survey: Manual and Interpretation Guide*. Boston MA: The Health Institute, New England Medical Center, 1993.

Ware JE, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36). I. Conceptual framework and item selection. *Med Care* 1992;30:473-483.

Watson DL, Tharp RG. Self-Directed Behavior: Self-Modification for Personal Adjustment (5th Ed.). Pacific Grove, California: Brooks/Cole, 1989.

Whelton PK, Appel LA, Espeland MA, Applegate WB, Ettinger WH, Kostis JB, Kumanyika S, Lacy CR, Johnson KC, Folmar S, Cutler JA. Sodium reduction and weight loss in the treatment of hypertension in older persons: A randomized Trial of Nonpharmacologic Interventions in the Elderly (TONE). *JAMA* 1998; 279:839-846.

Whelton PK, He J, Cutler JA, Brancati FL, Appel LJ, Follman D, Klag MJ. Effects of oral potassium on blood pressure. Meta-analysis of randomized controlled clinical trials. *JAMA* 1997; 227:1624-1632.

Whelton PK, Applegate WB, Ettinger WH, Espeland M, Kostis JB, Appel LJ, *et al.* Efficacy of weight loss and reduced sodium intake in the Trial of Nonpharmacologic Interventions in the Elderly (TONE). *Circulation* 1996; 94:I-178.

Working Group on Primary Prevention of Hypertension. *National High Blood Pressure Education Program: Working Group Report on Primary Prevention of Hypertension*. NIH Publication No. 93-2669; 1993.

Wright BM, Dore CF. A random-zero sphygmomanometer. *Lancet* 1970; 1:337-338.

Young DR, Haskell WL, Taylor CB, Fortmann SP. Effect of community health education on physical activity knowledge, attitudes, and behavior. The Stanford Five-City Project. *Am J Epidemiol* 1996; 144:264-274.

Zapka JG, Merriam P, Ockene J. Smoking cessation benefits in HMOs. *HMO Pract* 1997; 11:27-33.